CLINICAL TRIAL: NCT06851871
Title: A Phase 1, Open-label, Single-dose Study in Healthy Adult Participants to Assess the Bioequivalence Between Immediate Release Tablets and Minitablets, and to Assess the Food and pH Effect on the Pharmacokinetics of Deucravacitinib (BMS-986165) Administered as Minitablets
Brief Title: A Study to Evaluate the Bioequivalence Between Immediate Release Tablets and Minitablets of Deucravacitinib (BMS-986165), and the Effect of Food and pH on the Drug Levels of the Minitablets in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM011-1178
Record Dates: First submitted 2025-01-22; First posted 2025-02-28 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants
Keywords: Bioequivalence; Food Effect; pH Effect; Healthy Volunteers; Deucravacitinib
MeSH Terms: interventions — deucravacitinib; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BMS-986165 Formulation 1 (Experimental)
  Interventions: Drug: Deucravacitinib
- BMS-986165 Formulation 2 (Experimental)
  Interventions: Drug: Deucravacitinib
- BMS-986165 Formulation 2 + Fed (Experimental)
  Interventions: Drug: Deucravacitinib
- BMS-986165 Formulation 2 + Famotidine (Experimental)
  Interventions: Drug: Deucravacitinib; Drug: Famotidine

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
Drug: Famotidine — Specified dose on specified days
  Arms: BMS-986165 Formulation 2 + Famotidine

SUMMARY:
The purpose of this study is to evaluate the bioequivalence between immediate release tablets and minitablets of Deucravacitinib (BMS-986165), and the effect of food and pH on the drug levels of the minitablets in healthy adults.

ELIGIBILITY:
Inclusion Criteria

* Participants must be healthy as determined by no clinically significant deviation from normal in medical history, physical examination, vital signs, 12-lead ECGs, and clinical laboratory determinations in the opinion of the investigator.
* Participants must be willing and able to complete all study-specific procedures and visits.
* Participants must have a body mass index of 18.0 kg/m2 through 32.0 kg/m2, inclusive, and total body weight ≥ 50 kg (110 lb).

Exclusion Criteria

* Participants must not have any significant acute or chronic medical illness that presents a potential risk to the participant and/or may compromise the objectives of the study, including a history of/or acute liver disease in the opinion of the Investigator.
* Participants must not have evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, 12-lead ECG, or clinical laboratory determinations beyond what is consistent with the population reference ranges in the opinion of the investigator.
* Participants must not have any history of severe reaction to a drug (eg, anaphylactic, anaphylactoid, Stevens-Johnson, angioedematous), or adverse or allergic/hypersensitivity reaction to multiple drugs.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to day 20
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to day 20
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Up to day 20

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to day 44
Incidence of serious adverse events (SAEs) | Up to day 44
Incidence of AEs leading to discontinuation | Up to day 44
Number of participants with a clinically significant change from baseline in vital signs | Up to day 21
Number of participants with a change from baseline in 12-lead ECG results | Up to day 21
Number of participants with physical examination abnormalities | Up to day 21
  A physical examination includes the assessment of the following: head, eyes, ears, nose, and throat (HEENT), cardiovascular (including peripheral vascular), lungs, abdomen, dermatological, and a general neurological examination
Time of maximum observed plasma concentration (Tmax) | Up to day 20
Apparent terminal plasma half-life (T-HALF) | Up to day 20
Apparent total body clearance (CLT/F) | Up to day 20

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com